CLINICAL TRIAL: NCT05514197
Title: The Impact of Intravenous Vitamin C Combined With Nerve Blocks on Postoperative Pain and Recovery After Total Knee Arthroplasty.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chimei Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMMC11104/016
Record Dates: First submitted 2022-08-16; First posted 2022-08-24 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Ascorbic Acid; Postoperative Pain
Keywords: Ascorbic Acid; Total knee arthroplasty; Regional analgesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Ascorbic Acid; Tin Fluorides

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin C arm (Experimental): Intravenous loading of 100mg/kg ascorbic acid before induction, Maximus 10g
  Interventions: Drug: Ascorbic acid 100mg/kg, Maximus 10g
- Control arm (Placebo Comparator): Intravenous loading of the same volume Normal saline as experimental arm
  Interventions: Drug: Control Rx

INTERVENTIONS:
Drug: Ascorbic acid 100mg/kg, Maximus 10g — Intravenous loading of 100mg/kg ascorbic acid with normal saline, totally 100ml Completed before induction
  Arms: Vitamin C arm
Drug: Control Rx — Intravenous loading 100ml normal saline
  Arms: Control arm

SUMMARY:
The aim of this prospective randomized-control study was to evaluate the impact of a single high-dose intravenous vitamin C added to ultrasound-guided blocks at induction on postoperative pain, sngception and early functional rehabilitation of the knee joint in patients under-going total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

1. Physical status according to American Society of Anesthesiologists (ASA) I-III
2. Patients scheduled for total knee arthroplasty
3. Patients aged ranging from 50 to 80 years old

Exclusion Criteria:

1. Previous operation on the same knee
2. Allergy or intolerance to one of the study medications
3. Coagulopathy
4. Having lower limbs neuropathy
5. End-organ failure (CKD stage IV or V, NYHA III or IV)
6. BMI > 35
7. Chronic opioid use (>3 months) or drug abuser
8. Difficulty in communication (Impaired mental status)
9. Hyperuricemia or Glucose-6-phosphate dehydrogenase deficiency patient

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2024-01-11 (Actual)

PRIMARY OUTCOMES:
Numeric rating scale for pain | 15 minutes postoperatively
  11-point numeric scale ranges from '0' representing no pain to '10' representing the extreme pain
Numeric rating scale for pain | 1 hour postoperatively
  11-point numeric scale ranges from '0' representing no pain to '10' representing the extreme pain
Numeric rating scale for pain | 6 hours postoperatively
  11-point numeric scale ranges from '0' representing no pain to '10' representing the extreme pain
Numeric rating scale for pain | 24 hours postoperatively
  11-point numeric scale ranges from '0' representing no pain to '10' representing the extreme pain
Numeric rating scale for pain | 48 hours postoperatively
  11-point numeric scale ranges from '0' representing no pain to '10' representing the extreme pain
Numeric rating scale for soreness (Sngception) | 15 minutes after surgery
  11-point numeric scale ranges from '0' representing no soreness to '10' representing the extreme soreness
Numeric rating scale for soreness (Sngception) | 1 hours postoperatively
  11-point numeric scale ranges from '0' representing no soreness to '10' representing the extreme soreness
Numeric rating scale for soreness (Sngception) | 6 hours postoeratively
  11-point numeric scale ranges from '0' representing no soreness to '10' representing the extreme soreness
Numeric rating scale for soreness (Sngception) | 24 hours postoperatively
  11-point numeric scale ranges from '0' representing no soreness to '10' representing the extreme soreness
Numeric rating scale for soreness (Sngception) | 48 hours postoperatively
  11-point numeric scale ranges from '0' representing no soreness to '10' representing the extreme soreness

SECONDARY OUTCOMES:
Morphine consumption | 48 hours postoperatively
  Amount of IV morphine consumption postoperatively
Time to first rescue morphine requirement at post-anesthetic care unit | up to 2 hours
  Duration from arriving post-anesthetic care unit to requiring first morphine injection
Severity of postoperative nausea/ vomiting and dizziness | 48 hours postoperatively
  From 0 to 5, 0: non, 1: mild, 2: moderate, 3: severe, 4: unbearable

OTHER OUTCOMES:
Blood ascorbic acid concentration | Preoperative baseline and postoperative day1
  Blood ascorbic acid analysis
PostOP Knee joint range of motion | 72 hours postoperatively
  In degree from zero to 170

CONTACTS AND LOCATIONS:
Overall Officials: Jen-Yin Chen, Study Director — Department of Anesthesiology, Chimei Medical Center
Locations (1):
- Chi Mei Medical Center, Tainan, Tainan City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided